#### Official Title:

The Effect of Acceptance and Commitment Therapy—Based Psychoeducation on Self-Esteem and Interpersonal Problem-Solving Skills in Youth with Social Media Addiction

#### **Brief Title:**

ACT-Based Psychoeducation for Youth with Social Media Addiction

Acronym:

ACT-SM

#### **Institution:**

Kahramanmaraş Sütçü İmam University

## **Principal Investigator:**

Prof. Dr. Döndü Çuhadar

## Co-Investigator / Researcher:

Zeynep Kekeç, Research Assistant

# **Study Type:**

Interventional (Clinical Trial)

# Informed Voluntary Consent Form (For Adults)

(The form must be prepared in a way that is understandable to the volunteer, avoiding medical terminology and using plain language.)

#### Title of the Research

The Effect of Acceptance and Commitment Therapy-Based Psychoeducation on Self-Esteem and Interpersonal Problem-Solving Skills in Young People with Social Media Addiction

## The Purpose of the Research and Its Scientific Contributions

The aim of this study is to observe the effect of psychosocial education based on acceptance and commitment therapy, planned to address problems in the areas of self-esteem and interpersonal problem-solving skills, by identifying the effects of social media addiction, which is currently considered a behavioral disorder, on these areas. In this context, the aim is to reveal the relationship between the self-esteem and interpersonal problem-solving skills of young people addicted to social media and how these variables affect social media addiction, and to determine whether the psychoeducation application provides positive change in this area.

#### **Research Materials and Methods**

The study is a randomized controlled experimental study and will be conducted using a 2x3 split-plot design (experimental/control groups X pre-test/post-test/follow-up test).

University students who meet the research criteria and agree to participate will be administered the "Information Form," the "Rosenberg Self-Esteem Scale (RSES)," the "Social Media Addiction Scale-Adult Form (SMAS-AF)', and the 'Interpersonal Problem Solving Inventory' will be administered face-to-face by the researcher. Individuals with an item score average of 4 points or above on the Social Media Addiction Scale-Adult Form (SMAS-AF) will be included in the study.

# Biological Materials to be Collected from Volunteers and the Reason for Collection

#### The Reusability of Biological Materials

#### Procedures and/or Interventions to be Performed on Volunteers (Research Product/Method)

No action will be taken against the volunteer; training will be provided.

# Potential Risks and Harms to Volunteers

# Methods for Compensating for Risks and Losses Incurred

Circumstances Requiring Termination of the Volunteer's Participation in the Study
- Missing two consecutive sessions of training,

- Engaging in behavior that disrupts the group's order,
- Failing to comply with group rules,
- Not completing the assignments given during sessions.

#### **Responsibilities of Volunteers**

- Comply with psychoeducation rules,
- Comply with group rules
- Complete the assignments given during sessions.

#### **Insurance for Volunteers**

#### Payments to Volunteers

-

#### **Volunteer's Declaration**

I have carefully read and fully understood the above information. I have also been verbally informed by a researcher from the research team when necessary. It has been explained to me that my participation in the research is voluntary and that I may refuse to participate in the research or withdraw from it at any time without penalty or sanction and without losing any rights, and that records revealing my identity will be kept confidential, will not be disclosed to the public, and my identity will remain confidential even if the research results are published. Additionally, I have been informed that the ethics committee, institution, and other relevant health authorities may have direct access to my original medical records, but that this information will be kept confidential, and that by signing the written informed consent form, I or my legal representative will have

consented to such access. The research also specified the individuals I could contact to obtain further information about my rights or any adverse events related to the research, along with their 24-hour telephone numbers. I declare that I participated in the research entirely of my own free will and consent, and that no pressure was exerted on me to volunteer for the research.

| Volunteer | | | |
|------------|-----------|------|-------------|
| Name | Last name | Date | Signature |
| Researcher | | | |
| Name | Last name | | Phone |
| Zeynep | KEKEÇ | | 05452104507 |